CLINICAL TRIAL: NCT07360392
Title: Comparison of Postoperative Analgesic Effects of Two Different Anesthesia Techniques in Knee Arthroplasty: Nerve Blocks Named BiFeS and iPACK
Brief Title: BiFeS vs. iPACK in Postoperative Knee Arthroplasty Analgesia
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Amasya University (Other)
Responsible Party: Principal Investigator, Bülent Meriç Çam, Specialist Physician, Amasya University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2025-559
Record Dates: First submitted 2025-12-30; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Arthroplasty, Replacement, Knee; Pain, Postoperative; Anesthesia, Regional
Keywords: Pain Management; Knee Arthroplasty; BiFes; iPACK; Nerve Block
MeSH Terms: conditions — Pain, Postoperative; Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adductor Canal(ACB) + iPACK block (Active Comparator)
  Interventions: Procedure: Infiltration Between The Popliteal Artery and The Capsule of The Knee; Procedure: Adductor Canal Block
- Adductor Canal(ACB) + BiFeS block (Active Comparator)
  Interventions: Procedure: Biceps Femoris Short Head Block (BiFeS); Procedure: Adductor Canal Block

INTERVENTIONS:
Procedure: Biceps Femoris Short Head Block (BiFeS) — Under ultrasound guidance, the fascial plane between the short head of the biceps femoris and the semimembranosus muscles will be identified. The needle will be advanced into this plane using a lateral approach, and 20 mL of 0.25% bupivacaine will be injected. This injection area forms an anatomical corridor encompassing the terminal sensory branches of the common peroneal nerve, the popliteal extension of the posterior femoral cutaneous nerve, and the lateral genicular nerve branches. Thus, a broad sensory block is achieved along the posterolateral capsule of the knee without affecting motor fibers.
  Arms: Adductor Canal(ACB) + BiFeS block
Procedure: Infiltration Between The Popliteal Artery and The Capsule of The Knee — Under ultrasound guidance, the posterior aspect of the popliteal artery at the distal femur, at the level of the femoral condyles, will be targeted. The needle will be advanced using a medial approach, and 20 mL of 0.25% bupivacaine will be injected into the potential space between the artery and the posterior capsule of the knee. This technique blocks the terminal genicular nerve branches innervating the posterior capsule while sparing motor fibers.
  Arms: Adductor Canal(ACB) + iPACK block
Procedure: Adductor Canal Block — The block will be performed under ultrasound guidance at the distal femoral triangle, just below the apex of the femoral triangle. This level lies deep to the sartorius muscle and represents the lower boundary of the vastoadductor membrane and the beginning of the adductor canal. The ultrasound probe will be placed transversely on the medial thigh to visualize the femoral artery, and the saphenous nerve running lateral to the artery will be targeted. A total of 20 mL of 0.25% bupivacaine will be slowly injected beneath the sartorius muscle and lateral to the femoral artery to allow spread along the adductor canal. This injection at this level affects both the saphenous nerve and the motor branch of the vastus medialis, providing an effective sensory block of the anterior and medial aspects of the knee joint.

SUMMARY:
The Biceps Femoris Short Head (BiFeS) block is a new fascial plane block technique targeting the sensory innervation of the posterolateral capsule of the knee while preserving motor function. The aim of this study is to evaluate the postoperative analgesic efficacy of the BiFeS block combined with the adductor canal block (ACB) in patients undergoing total knee arthroplasty, compared to ACB + iPACK block. The study is planned as a prospective, randomized, double-blind, parallel two-group trial. Patients will be randomized in a 1:1 ratio to receive ACB + iPACK (Group A) or ACB + BiFeS (Group B). Postoperative pain scores (VAS), opioid consumption, early mobilization, and quality of recovery (QoR-15) outcomes will be compared.

DETAILED DESCRIPTION:
Total knee arthroplasty (TKA) is an effective surgical method for the treatment of advanced osteoarthritis, reducing pain and improving functional capacity. However, approximately 30-40% of cases experience severe postoperative pain, and 20-31% of patients develop persistent postoperative pain (1, 2). This not only delays early mobilization and rehabilitation but also negatively affects patient satisfaction and overall recovery.

Enhanced Recovery After Surgery (ERAS) protocols emphasize that effective postoperative analgesia is indispensable for early mobilization and functional recovery. Multimodal analgesic strategies, particularly combinations of motor-sparing regional anesthesia techniques, are a cornerstone of these protocols (3).

One of these regional anesthesia techniques, the femoral nerve block (FNB), provides strong analgesic efficacy but reduces quadriceps strength, increasing the risk of falls. Therefore, in recent years, "motor-sparing" approaches aimed at preserving motor function have gained prominence (4).

Recent high-level network meta-analyses have shown that combinations of motor-sparing regional techniques provide superior outcomes compared to single blocks. In a 2024 meta-analysis by Wang et al., including 30 randomized controlled trials (RCTs), the combination of continuous adductor canal block (cACB) + genicular nerve block (GNB) among motor-sparing approaches provided the lowest rest pain scores at 24 and 48 hours, while cACB + iPACK + GNB combination most effectively reduced pain on movement (5). In the same study, this combination also demonstrated the highest performance in functional recovery indicators, with the shortest Timed-Up-and-Go (TUG) time and greatest range of motion.

Similarly, a 2025 Bayesian network meta-analysis by Migliorini et al., analyzing 77 RCTs, reported the lowest visual analog scale (VAS) scores between postoperative days 1-3 with continuous periarticular analgesia/local infiltration analgesia (PCI/LIA); this was followed by continuous FNB/PCI and continuous ACB applications, respectively (6).

Both analyses emphasized that multimodal approaches, particularly combinations of ACB, iPACK, GNB, or LIA, reduce opioid consumption and support early mobilization.

Another large-scale Bayesian network meta-analysis published by Xue et al. in 2024 reported that the ACB + iPACK combination significantly reduced pain at rest and on movement at 48 hours compared to single blocks (ACB, FNB, GNB, iPACK), decreased opioid consumption, and accelerated early mobilization (7).

However, current techniques have several limitations. LIA is surgeon-dependent, requires a large local anesthetic volume (100-150 mL), and shows variable efficacy due to a lack of standardization in composition/concentration. High volumes also increase the risk of local anesthetic systemic toxicity (LAST). While FNB provides effective pain control, it is not compatible with motor-sparing goals due to quadriceps weakness. Continuous blocks offer analgesic advantages but add logistical burdens due to the need for catheters, pumps, and monitoring.

In this context, new regional techniques are needed that preserve motor function while targeting the sensory innervation of the posterolateral capsule. To address this, the Biceps Femoris Short Head (BiFeS) block, introduced by Kılıçaslan et al. in 2025, is an innovative fascial plane block technique targeting the nerve branches innervating the posterolateral capsule of the knee (8). Ultrasound-guided injection between the short head of the biceps femoris and semimembranosus muscles allows the spread of local anesthetic along the natural fascial plane between these two muscles. This plane constitutes an anatomical corridor including the terminal sensory branches of the common peroneal nerve, the popliteal extension of the posterior femoral cutaneous nerve, and lateral genicular nerve branches. The oblique orientation of muscle fibers facilitates proximal and distal spread of the local anesthetic, creating a broader sensory block encompassing the posterolateral capsule of the knee. Thus, the BiFeS block is expected to provide a wider sensory area than the iPACK block without affecting motor fibers.

Cadaveric studies and early clinical data suggest that the BiFeS block combined with ACB may contribute to multimodal approaches by enhancing postoperative analgesia while preserving motor-sparing efficacy (8). However, no randomized controlled trial has yet demonstrated the clinical effectiveness of this technique.

The hypothesis of this study is that the BiFeS block applied in combination with ACB provides superior postoperative analgesia compared to the iPACK block applied with ACB.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral total knee arthroplasty
* Classified as ASA physical status I-III

Exclusion Criteria:

* Scheduled for revision arthroplasty or bilateral surgery
* Allergy to local anesthetics or contraindication to regional blocks
* Neurological disorders, peripheral neuropathy, or conditions affecting lower extremity muscle strength
* Coagulopathy or receiving anticoagulant therapy
* History of severe liver, kidney, or heart failure
* Chronic opioid use or history of substance abuse
* Patients experiencing intraoperative complications (e.g., excessive bleeding)
* Cases in which adequate sensory blockade is not achieved after the block

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
Postoperative 12th hour pain score | Postoperative 12th hour
  Postoperative 12th hour pain score (will be evaluated with Visuel Analog Scale) Higher scores indicate worse condition

SECONDARY OUTCOMES:
Postoperative Rest and Movement VAS Scores at 2, 4, 6, 8, 12, 24, 48, 72 Hours and 1, 3 Months | Postoperative 1st, 2nd, 4th, 8th, 12th, 16th, 24th, 48th hours and 1st ,3th Months
  Higher scores indicate worse condition
Time to Postoperative Rescue Analgesia (minutes) | Postoperative 72th hours
  Time to Postoperative Rescue Analgesia (minutes; longer duration indicates slower attainment of VAS score of 4, with higher scores reflecting better analgesia)
Postoperative Cumulative Tramadol Consumption (mg) | Postoperative 72th hours
Postoperative Complications such as Nausea and Vomiting | Every 12 hours during the first 72hours postoperative hours
Quality of Recovery-15 (QoR-15) Score | preoperative day 1 and postoperative day 1
  It is a test used to assess postoperative recovery quality.The Quality of Recovery-15 (QoR-15) scale has a minimum score of 0 and a maximum score of 150, with higher scores indicating better postoperative recovery and lower scores indicating poorer recovery
Time to Meet Physiotherapy Criteria for Hospital Discharge | Every 12 hours during the first 72hours postoperative hours
  Ability to walk independently from bed to bathroom, walk in the corridor without a walker, and sit down and stand up from a chair independently

CONTACTS AND LOCATIONS:
Locations (1):
- Amasya University Sabuncuoğlu Şerefeddin Training and Research Hospital, Amasya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No